CLINICAL TRIAL: NCT00213759
Title: Prevention Trial of Nosocomial Infections in Neutropenic Prematures With G-CSF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2712; 0203222
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Neutropenia in Prematures
Keywords: neutropenia; prematurity; nosocomial infection; G-CSF
MeSH Terms: conditions — Neutropenia; Premature Birth; Cross Infection | interventions — Filgrastim

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- groupe filigrastin (Active Comparator)
  Interventions: Drug: filgrastim
- groupe placebo (Placebo Comparator)
  Interventions: Drug: dextrose 5%

INTERVENTIONS:
Drug: filgrastim — The G-CSF (filigrastin) will be administered by intravenous way with the amount of 10 µg/kg/day during 3 days . The infusion will last from 20 to 40 minutes according to weight of the child and the product will be diluted in dextrose 5%.
  Arms: groupe filigrastin
Drug: dextrose 5% — The placebo (dextrose 5% ) will be injected by intravenous way with the amount of 0.66 ml/kg during 3 days consecutive. The infusion will last from 20 to 40 minutes.
  Arms: groupe placebo

SUMMARY:
Prevention trial of nosocomial infections in neutropenic prematures with G-CSF

ELIGIBILITY:
Inclusion Criteria:

< 33 weeks GA neutropenic during at least 24 hours in the first 3 weeks of life and not infected at time of inclusion < 35 if birth weight < 1500 g

Ages: 2 Days to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2002-03; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
survival without infection at 4 weeks after treatment | one month

SECONDARY OUTCOMES:
survival free of infection at 2 weeks after treatment,mortality, increase of neutrophile, number of septic event, incidence of chronic lung disease, necrotizing enterocolitis, cerebral us abnormalities, retinopathy , duration of hospitalisation stay | one month

CONTACTS AND LOCATIONS:
Overall Officials: Jean Messer, MD, Principal Investigator — Hopitaux Universitaires de Strasbourg
Locations (9):
- France (9):
  - Xavier Hernandorena, Bayonne
  - Alain Menget, Besançon
  - Jean-Louis Demarquez, Bordeaux
  - Bernard Guillois, Caen
  - Marie Thieuleux, Calais
  - André Labbe, Clermont-Ferrand
  - Jean-Bernard Gouyon, Dijon
  - Pierre Andrini, Grenoble
  - Jean Messer, Strasbourg

REFERENCES:
- [Derived] Kuhn P, Messer J, Paupe A, Espagne S, Kacet N, Mouchnino G, Klosowski S, Krim G, Lescure S, Le Bouedec S, Meyer P, Astruc D. A multicenter, randomized, placebo-controlled trial of prophylactic recombinant granulocyte-colony stimulating factor in preterm neonates with neutropenia. J Pediatr. 2009 Sep;155(3):324-30.e1. doi: 10.1016/j.jpeds.2009.03.019. Epub 2009 May 24. PMID 19467544